CLINICAL TRIAL: NCT06862752
Title: Bilateral Ultrasound-Guided Erector Spinae Plane Block or Serratus Anterior Plane Block For Postoperative Analgesia in Breast Reduction Surgery: A Prospective, Randomized and Controlled Trial
Brief Title: Erector Spinae Plane Block Versus Serratus Anterior Plane Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Leyla Kılınc, associate professor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: leyla-25
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Post Operative Pain; Opioid-Related Disorders
Keywords: post operative pain; opioid consumption; erector spinae block; serratus anterior plane block
MeSH Terms: conditions — Pain, Postoperative; Opioid-Related Disorders | interventions — Parapsychology; Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP block group (Active Comparator): Bilateral ultrasound guided erector spine plane (ESP) block will be performe preoperatively at T5 level. 20 mL local anesthetics (10 mL 0.5% bupivacaine + 10 mL serum physiologic % l) will be injected deep to the erector spinae muscle
  Interventions: Procedure: erector spine plane (ESP) block
- SAP Block grup (Other): Bilateral ultrasound guided serratus plane block with 20 ml %0,25 bupivacaine at the midaxillary 5. Rib
  Interventions: Procedure: Serratus Anterior Plane Block

INTERVENTIONS:
Procedure: erector spine plane (ESP) block — Bilateral ultrasound guided erector spine plane (ESP) block will be performe preoperatively at T5 level. 20 mL local anesthetics (10 mL 0.5% bupivacaine + 10 mL serum physiologic % l) will be injected deep to the erector spinae muscle.
  Arms: ESP block group
Procedure: Serratus Anterior Plane Block — Bilateral ultrasound guided serratus plane block with 20 ml %0,25 bupivacaine at the midaxillary 5. Rib
  Arms: SAP Block grup

SUMMARY:
the aim of the study compare the analgesic effect of erector spinae block and serratus anterior block in breast surgery

DETAILED DESCRIPTION:
Breast reduction surgery is a common cosmetic surgical procedure. Providing effective analgesia has a crucial role in reducing side effects, catalyzing postoperative recovery, and increasing patient satisfaction. Regional anesthesia techniques are generally used for postoperative analgesia to decrease opioid-related side effects. Fascial plane block has gained popularity for breast analgesia. The investigator aimed to consider the effects of ESP block or Serratus Anterior Plane block on postoperative analgesia in breast reduction surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I-II,
* 18-65 years of age, adult,
* female patients
* undergoing elective breast reduction surgery

Exclusion Criteria:

* Allergy to amide-type local anesthetics
* Infection at the block injection site
* Severe obesity (BMI > 35 kg/m2)
* Liver or renal deficiency
* Patients with anatomical deformities
* Recent use of analgesic drugs
* Patient refusal or inability to consent

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 24 hour
  Tramadol consumption in Patient Controlled Analgesia device postoperative 24 hours.

SECONDARY OUTCOMES:
Pain assessed by NRS | 24 hour
  Post operative pain will be evaluated with Numeric rating scale (NRS) score of 0-10 (0= no pain and 10= pain) and will be recorded at 0,1,4,12,24. At hours postoperatively.
Rate of opioid related side effects | 24 hour
  Opioid related side effects such as nause/vomiting, pruritis, bradycardia, hypotension will be evaluated at intervals up to 24 hours.
Blooad loss | during surgery
  Peroperative and postoperative blood loss and amaoun of eritrosit suspansion
Remifentanil consumption | during surgery
  Peroperative Remifentanil consumption
Length of stay in hospital | 30 days
  Length of stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: AYSE SURHAN CINAR, Study Chair — SISLI HAMIDIYE ETFAL RESEARCH AND TRAINING
Locations (1):
- Sisli etfal research and training hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No